CLINICAL TRIAL: NCT06835140
Title: CD123-Targeted CD16 Antibody-Modified NK Cell Immunotherapy for Refractory/Relapsed Acute Myeloid Leukemia (R/R AML)
Brief Title: CD123-CD16-NK Cells Immunotherapy for AML
Acronym: CD123-CD16-NK
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chunji Gao (Other)
Collaborators: Chinese PLA General Hospital (Other)
Responsible Party: Sponsor-Investigator, Chunji Gao, Principal Investigator, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2024-653-01
Record Dates: First submitted 2025-01-07; First posted 2025-02-19 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: AML (Acute Myelogenous Leukemia); NK Cell; CD123+ Acute Myeloid Leukemia
Keywords: CD123-CD16 bispecific antibody; NK cell; Refractory/relapsed AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CD123-CD16 bispecific antibody-modified NK cells for the treatment of CD123-positive R/R AML (Experimental): Patients scheduled to receive CD123-CD16-NK cell infusions undergo lymphocyte-depleting chemotherapy from day -5 to day -3. After completing preconditioning, 48 hours later, patients are intravenously infused with NK cells at a dose of 1×10⁷ cells/kg (100-150 ml volume) within 10 to 15 minutes. Infusions are administered every 96-120 hours for a total of three times. Subsequently, patients receive escalating NK cell doses of 2×10⁷ cells/kg and 4×10⁷ cells/kg. Vital signs (temperature, heart rate, respiratory rate, blood pressure, etc.) are monitored before and after infusion. Baseline data during NK cell infusion are also recorded. For each dose group, only one patient initially receives a single NK cell infusion, followed by a 3-day observation period to ensure safety before proceeding with a second infusion. If no adverse events occur in the initial dose group, the next dose group is infused accordingly, and the process continues similarly.
  Interventions: Drug: Donor-derived CD123-CD16 bispecific antibody-modified NK cells

INTERVENTIONS:
Drug: Donor-derived CD123-CD16 bispecific antibody-modified NK cells — Patients enrolled sequentially received varying doses of NK cell infusions. The first three patients received 1×10⁷ cells/kg, the next three received 2×10⁷ cells/kg, and the final three received 4×10⁷ cells/kg.

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of CD123-CD16 bispecific antibody-modified NK cells in treating patients with CD123-positive relapsed or refractory Acute Myeloid Leukemia (RR AML). It will also assess the safety of this modified NK cell therapy.

The main questions： Does the infusion of CD123-CD16 bispecific antibody-modified NK cells induce remission in RR AML patients? What are the safety and potential adverse effects associated with the administration of these modified NK cells? Researchers will administer CD123-CD16 bispecific antibody-modified NK cells to RR AML patients and compare the outcomes to existing treatment options to determine efficacy and safety.

Participants will:

Undergo lymphocyte-depleting chemotherapy Fludarabine&Cyclophosphamide from day -5 to day -3 before NK cell infusion.

Receive intravenous infusions of modified NK cells at escalating doses:

The first three patients will receive 1×10⁷ cells/kg. The next three patients will receive 2×10⁷ cells/kg. The final three patients will receive 4×10⁷ cells/kg. Have NK cell infusions administered every 96-120 hours for a total of three infusions, with each infusion completed within 10 to 15 minutes.

Undergo dose escalation with subsequent groups only after confirming the safety of the previous dose group.

Have their vital signs (temperature, heart rate, respiratory rate, blood pressure, etc.) monitored before and after each infusion.

Keep baseline data records during NK cell infusions. Participate in follow-up assessments to monitor disease remission and detect any adverse events.

This trial aims to provide new treatment options for RR AML patients by leveraging the targeted cytotoxic effects of CD123-CD16 bispecific antibody-modified NK cells to achieve disease remission.

ELIGIBILITY:
Inclusion Criteria:

1. Age: Between18 years and 70 years.
2. Diagnosis and Treatment History:

   Diagnosed with Acute Myeloid Leukemia (AML) in the hospital. Has undergone multiple first-line clinical treatments and has developed resistance to current treatments. Relapse after original induction therapy failure with a predicted survival of more than three months.
3. CD123 Expression:

   Flow cytometry detection shows CD123-positive AML cells.CD123 expression level is not less than 20%.
4. Hospital Examination Criteria:
5. Performance Status:

   ECOG Performance Status score of 0-2 or Karnofsky Performance Status (KPS) score greater than 80.
6. Donor Availability:
7. Have a suitable healthy donor and agree to peripheral blood collection.

Exclusion Criteria:

1. Specific AML Subtype:

   Diagnosed with Acute Promyelocytic Leukemia(APL).
2. CD123 Expression:

   Flow cytometry shows CD123 negative or CD123 expression level less than 20%.
3. Prior Treatment Toxicity:

   Persistent non-hematologic toxicity of grade 2 or higher related to previous treatments.
4. GVHD Requiring Immunosuppression:

   Patients requiring immunosuppressants for grade II-IV acute Graft-Versus-Host Disease (GVHD).
5. Recent Steroid Treatment:

   Systemic steroid treatment within 7 days prior to first study drug treatment (excluding topical and inhaled corticosteroids or short-term prophylactic steroid treatment).
6. Severe Cardiovascular and Cerebrovascular Diseases:

   Certain cardiovascular and cerebrovascular diseases within 6 months prior to first dose.

   New York Heart Association (NYHA) classification ≥3 or uncontrolled malignant arrhythmias.Other cardiovascular and cerebrovascular diseases deemed unsuitable by the investigator.
7. Pregnancy and Lactation:

   Pregnant or breastfeeding women (the safety of this treatment for unborn babies is unknown).

   For female participants, pregnancy must be confirmed negative by serum or urine pregnancy test within 48 hours before infusion.
8. Infections:

   Active Hepatitis B,Hepatitis C virus infection, Peripheral blood CMV-DNA ≥500 copies/mL, HIV/AIDS infection and any uncontrolled active infection.
9. Allergic Reactions:

   Allergic to immunotherapy and related drugs.
10. Neurological Diseases:

Neurological diseases such as neurodegenerative diseases, primary central nervous system tumors/infections, multiple sclerosis, epilepsy, severe peripheral neuropathy, etc.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-02-21 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | Bone marrow aspiration assessments are conducted one week after each patient's treatment completion, followed by evaluations at 1 month, 3 months, and 6 months.
  Overall Response Rate
CR | Bone marrow aspiration assessments are conducted one week after each patient's treatment completion, followed by evaluations at 1 month, 3 months, and 6 months.
  Complete Remission Rate
AE | 14 days-28 days after infusion
  Adverse events related to cell reinfusion (≥ Grade 3 treatment-related organ toxicity, laboratory tests, and Grade 4 hematologic toxicity, etc.) and number of participants with treatment-related AEs assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Progressive Disease (PD) | 14 days-28 days after infusion
  PD parameters: content of CD123+AML cells in peripheral blood ; plasma cytokine levels at various time points;
Stable Disease (SD) | 14 days-28 days after infusion
  the condition without significant progression nor significant reduction in AML cells after treatment. The disease is stable, with no significant change in the number of leukemia cells in peripheral blood or bone marrow assessed by IRC.
Progression-free survival (PFS) | through study completion, an average of 6-12moths
  the time from cell last infusion to the first assessment of tumor progression, relapse, or death for any reason
Overall survival (OS) | through study completion, an average of 6-12moths
  the time from cell last infusion to death for any reason

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, China, China

IPD SHARING:
Plan to Share IPD: No